CLINICAL TRIAL: NCT04497558
Title: The Clinical Efficiency of Transcriptome-based Endometrial Receptivity Assessment (Tb-ERA) in Chinese Patients With Recurrent Implantation Failure (RIF)
Brief Title: The Clinical Efficiency of Tb-ERA in Chinese RIF Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ShangHai Ji Ai Genetics & IVF Institute (Other)
Responsible Party: Principal Investigator, Wenbi Zhang, Clinical Professor, ShangHai Ji Ai Genetics & IVF Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: JIAI 2020-07
Record Dates: First submitted 2020-07-28; First posted 2020-08-04 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Endometrial Receptivity; Repeated Implantation Failure
Keywords: endometrial receptivity array; Repeated implantation failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERA group (Experimental): In the experimental group, those patients undergo endometrial receptivity array. According to the results of endometrial receptivity array, the transplantation time will be adjusted and retransplantation will be carried out.
  Interventions: Diagnostic Test: Endometrium biopsy
- Control group (No Intervention): In the control group, those patients do not receive any treatment before next cycle of transfer. In the control group, no intervention will be performed.

INTERVENTIONS:
Diagnostic Test: Endometrium biopsy — In the experimental group, those patients undergo endometrial receptivity array. In the control group, those patients do not receive any treatment before next cycle of transfer. In the experimental group, according to the results of endometrial receptivity array, the transplantation time will be adjusted and retransplantation will be carried out. In the control group, no intervention will be performed.
  Arms: ERA group

SUMMARY:
In order to further explore the clinical utility of endometrial receptivity array in patients with repeated implantation failure, the patients divide into the experimental group or the control group. In the experimental group, those patients undergo endometrial receptivity array. In the control group, those patients do not receive any treatment before next cycle of transfer. In the experimental group, according to the results of endometrial receptivity array, the transplantation time will be adjusted and retransplantation will be carried out. Statistical analysis of the two groups of primary endpoint and secondary endpoint are done.

DETAILED DESCRIPTION:
In the field of assisted reproduction techonology, there are still 10% of patients with repeated implantation failure. In order to further explore the clinical utility of endometrial receptivity array in patients with repeated implantation failure, the patients divide into the experimental group or the control group. In the experimental group, those patients undergo endometrial receptivity array. In the control group, those patients do not receive any treatment before next cycle of transfer. In the experimental group, according to the results of endometrial receptivity array, the transplantation time will be adjusted and retransplantation will be carried out. In the control group, no intervention will be performed. Statistical analysis of the two groups of primary endpoint (clinical pregnancy rate) and secondary endpoint (endometrial implantation window evaluation results, embryo implantation rate, biochemical pregnancy rate, early abortion rate, ectopic pregnancy rate) are done. Through the comparative analysis of clinical outcomes to verify the clinical efficacy of endometrial receptivity analysis in patients with repeated implant failure, this method will provide a new treatment for repeated implant failure population.

ELIGIBILITY:
Inclusion Criteria:

1. People with unexplained repeated implantation failure (3 or more times of transplantation, at least 4 or more high-quality embryos failed to conceive).
2. Age: 20-40 years old.
3. BMI: 19 - 24.
4. The thickness of endometrium is more than or equal to 7 mm.

Exclusion Criteria:

1. Known causes of embryo implantation failure, such as infection, reproductive tract malformation, uterine cavity factors, immune factors, hydrosalpinx, etc.
2. Decreased ovarian function (meet the following at least two criteria: ① 10u / L < basal follicle stimulating hormone (FSH) < 25U / L, and / or estradiol (E2) > 292.8pmol/l, and / or FSH / LH > 3; ② the number of antral follicles < 5-7 on the second to third day of menstruation; and (or) antimullerian hormone (AMH) < 0.5-1.1ng/ml.
3. People with genetic history.
4. Those who have done abortion and the histogenetic analysis are positive.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 6 months
  Clinical pregnancy rate in patients

SECONDARY OUTCOMES:
Endometrial implantation window evaluation results | 6 months
  Endometrial implantation window evaluation results in tested patients
Embryo implantation rate | 6 months
  Embryo implantation rate in patients
Biochemical pregnancy rate | 6 months
  Biochemical pregnancy rate in patients
Early abortion rate | 6 months
  Early abortion rate in patients
Ectopic pregnancy rate | 6 months
  Ectopic pregnancy rate in patients

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxi Sun, Study Chair — Obstetrics and Gynecology Hospital affiliated to Fudan University
Locations (1):
- Shanghai Ji Ai Genetics & IVF Institute, Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruiz-Alonso M, Blesa D, Diaz-Gimeno P, Gomez E, Fernandez-Sanchez M, Carranza F, Carrera J, Vilella F, Pellicer A, Simon C. The endometrial receptivity array for diagnosis and personalized embryo transfer as a treatment for patients with repeated implantation failure. Fertil Steril. 2013 Sep;100(3):818-24. doi: 10.1016/j.fertnstert.2013.05.004. Epub 2013 Jun 4. PMID 23756099
- [Background] Hashimoto T, Koizumi M, Doshida M, Toya M, Sagara E, Oka N, Nakajo Y, Aono N, Igarashi H, Kyono K. Efficacy of the endometrial receptivity array for repeated implantation failure in Japan: A retrospective, two-centers study. Reprod Med Biol. 2017 Jun 27;16(3):290-296. doi: 10.1002/rmb2.12041. eCollection 2017 Jul. PMID 29259480
- [Derived] Zhang WB, Li H, Lu X, Chen JL, Li L, Chen JC, Wu H, Sun XX. The clinical efficiency of transcriptome-based endometrial receptivity assessment (Tb-ERA) in Chinese patients with recurrent implantation failure (RIF): A study protocol for a prospective randomized controlled trial. Contemp Clin Trials Commun. 2022 May 28;28:100928. doi: 10.1016/j.conctc.2022.100928. eCollection 2022 Aug. PMID 35669489